CLINICAL TRIAL: NCT06895733
Title: A Multi Cohort Phase IB/II Clinical Study of Pazopanib Combined With Palbociclib for Third Line and Beyond Treatment of Refractory Solid Tumors With Co-amplified in the 11q13(FGF3/4/19/CCND1)
Brief Title: Study of Pazopanib Combined With Palbociclib for Refractory Solid Tumors With Co-amplified in the 11q13(FGF3/4/19/CCND1)
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Tianjin Medical University Second Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MyCustom-Basket trials-PaPa
Record Dates: First submitted 2025-03-18; First posted 2025-03-26 (Actual); Last update posted 2025-03-26 (Actual); Status verified 2025-03

CONDITIONS: Solid Tumor, Adult; Next-generation Sequencing; Precision Medicine
MeSH Terms: interventions — pazopanib; palbociclib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Uroepithelial carcinoma (Experimental): Uroepithelial carcinoma with co-amplification of 11q13 region(FGF3/4/19/CCND1) or FGFR1/FGFR2 amplification
  Interventions: Drug: Pazopanib Oral Tablet; Drug: Palbociclib
- Head and neck squamous cell carcinoma (Experimental): Head and neck squamous cell carcinoma co-amplified in the 11q13 region(FGF3/4/19/CCND1)
  Interventions: Drug: Pazopanib Oral Tablet; Drug: Palbociclib
- Other solid carcinoma (Experimental): Other solid carcinoma co-amplified in the 11q13 region(FGF3/4/19/CCND1)
  Interventions: Drug: Pazopanib Oral Tablet; Drug: Palbociclib

INTERVENTIONS:
Drug: Pazopanib Oral Tablet — Orally administered once daily (100mg)for 21 consecutive days, followed by a 7-day cessation of medication; Every 28 days is a treatment cycle.
Drug: Palbociclib — Oral treatment once a day, with a cycle of 28 days. In the safety introduction section, the initial dose of pazopanib is 400mg, and in the dose escalation queue, the dose of pazopanib is 600mg.

SUMMARY:
The efficacy and safety of Pazopanib combined with Palbociclib in the third line and above treatment of refractory solid tumors co amplified in the 11q13 region (FGF3/4/19/CCND1).

DETAILED DESCRIPTION:
Based on literature review, this study first conducted a phase Ib study to observe the dose limiting toxicity (DLTs) of the combination therapy of pazopanib and palbociclib and to determine the recommended dose for phase II study (RP2D); Further phase II studies will be conducted to evaluate the efficacy of pazopanib combined with palbociclib in the third line and above treatment of refractory solid tumors co amplified in the 11q13 region using objective response rate (ORR) or progression free survival 2/progression free survival 1 (PFS2/PFS1). And observe and evaluate the progression free survival (PFS), time to remission (TTR), disease control rate (DCR), and overall survival (OS) of pazopanib combined with palbociclib for third line and above treatment of refractory solid tumors co amplified in the 11q13 region. Evaluate the safety of Pazopanib combined with palbociclib for the third line and above treatment of refractory solid tumors co amplified in the 11q13 region.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntarily join this study and sign an informed consent form;
2. ≥ 18 years old;
3. Patients with metastatic solid tumors diagnosed by histology or cytology; Queue 1:11q13 co amplified or FGFR1/FGFR2 amplified urothelial carcinoma Queue 2: Head and neck squamous cell carcinoma co amplified in 11q13 region Queue 3:11q13 co amplified other solid tumors
4. Disease progression or intolerable toxicity confirmed by imaging during or after treatment with at least two standard treatment regimens in the past;
5. According to RECIST 1.1, there must be at least one measurable lesion;
6. Can swallow pills normally;
7. ECOG score: 0-2;
8. Expected survival period ≥ 12 weeks;
9. The function of important organs meets the following requirements (no blood components or cell growth factor drugs are allowed to be used within 14 days before the first medication):

   Absolute neutrophil count ≥ 1.5 × 109/L; Platelets ≥ 100 × 109/L; Hemoglobin ≥ 90 g/L; Serum albumin ≥ 30 g/L; Serum total bilirubin ≤ 1.5 × ULN; ALT and AST ≤ 2.5 × ULN, and if there is liver metastasis, ALT and AST ≤ 5ULN; AKP≤ 2.5×ULN；Serum creatinine ≤ 1.5 × ULN; International normalized ratio (INR) ≤ 1.5 (not receiving anticoagulant therapy);
10. Non surgical sterilization or female patients of childbearing age are required to use a medically approved contraceptive measure (such as intrauterine device, contraceptive pill, or condom) during the study treatment period and within 3 months after the end of the study treatment period; Female patients of childbearing age who undergo non-surgical sterilization must have a negative serum or urine HCG test within 7 days prior to their first medication; And it must be during non lactation period; For male patients whose partners are women of childbearing age, effective contraception methods should be used during the trial period and within 3 months after the last administration of the trial drug.

Exclusion Criteria:

1. Known history or evidence of interstitial lung disease or active non infectious pneumonia;
2. Known to have central nervous system metastases;
3. Within the past 5 years or simultaneously with other malignant tumors (excluding cured skin basal cell carcinoma and cervical carcinoma in situ);
4. Suffering from hypertension and unable to achieve good control with antihypertensive medication (systolic blood pressure ≥ 140 mmHg or diastolic blood pressure ≥ 90 mmHg); Allow the above parameters to be achieved through the use of antihypertensive therapy; Previously experienced hypertensive crisis or hypertensive encephalopathy;
5. There are uncontrolled clinical symptoms or diseases of the heart, such as: (1) NYHA grade 2 or above heart failure, (2) unstable angina pectoris, (3) myocardial infarction within 1 year, (4) clinically significant supraventricular or ventricular arrhythmias requiring treatment or intervention, (5) QTc>450ms (male); QTc>470ms (female);
6. For those undergoing thrombolytic or anticoagulant therapy, prophylactic use of low-dose aspirin and low molecular weight heparin is allowed;
7. Within the first 3 months of enrollment, there have been significant clinical bleeding symptoms or clear bleeding tendencies; If fecal occult blood is positive during the baseline period, a follow-up examination can be conducted. If the result is still positive after the follow-up examination, gastroscopy examination is required;
8. Tumor invasion of important blood vessels, or the possibility of tumor invasion of important blood vessels in the future research period determined by imaging, may lead to fatal bleeding;
9. If the patient has pleural effusion, ascites, or pericardial effusion that requires drainage, and the researcher evaluates the symptoms to be stable after drainage, they can be enrolled;
10. Occurrence of arterial/venous thrombosis events within the first 6 months of enrollment, such as cerebrovascular accidents (including temporary ischemic attacks, cerebral hemorrhage, cerebral infarction), deep vein thrombosis, and pulmonary embolism;
11. Known genetic or acquired bleeding and thrombophilia tendencies (such as in hemophilia patients, coagulation dysfunction, etc.);
12. Within 6 months prior to the start of treatment, there has been an abdominal fistula, gastrointestinal perforation, or abdominal abscess;
13. Significant vascular disease (such as aortic aneurysm requiring surgical repair or recent peripheral arterial thrombosis) occurred within 6 months prior to the start of the study treatment;
14. Severe, unhealed, or cracked wounds, as well as active ulcers or untreated fractures;
15. Received major surgical treatment (excluding diagnosis) within 4 weeks before the start of the study treatment or expected to undergo major surgical treatment during the study period;
16. Urine routine shows that urine protein is ≥++and has been confirmed to have a 24-hour urine protein level>1.0 g;
17. Previously received radiotherapy (excluding palliative radiotherapy for bone lesions), chemotherapy, surgery (excluding biopsy), and less than 4 weeks before the first study medication after completion of treatment (last medication); The last dose of antibody administration is less than 4 weeks after the first study medication; Molecular targeted therapy (including other oral targeted drugs used in clinical trials) for patients with less than 5 drug half lives from the first study drug, or adverse reactions caused by previous treatment (excluding hair loss) that have not recovered to ≤ CTCAE grade 1;
18. Suffering from active infection, having unexplained fever ≥ 38.5 ℃ within 7 days before medication, or baseline white blood cell count>15 × 109/L;
19. Suffering from congenital or acquired immune dysfunction (such as HIV infected individuals); Hepatitis B surface antigen (HBsAg) positive and hepatitis B virus deoxyribonucleic acid (HBV DNA) ≥ 2000 IU/ml, or hepatitis C virus antibody positive;
20. Previously received anti angiogenic therapy;
21. According to the researchers' judgment, the patient may have other factors that may affect the research results or cause the study to be terminated midway, such as alcohol abuse, drug abuse, other serious illnesses (including mental illnesses) that require concomitant treatment, serious laboratory test abnormalities, and family or social factors that may affect the patient's safety.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Estimated)
Dates: Start 2024-11-27 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) | Through study completion, an expected average of 1 year.
  Objective Response Rate (ORR) assessed according to the evaluation criteria for the efficacy of solid tumors (RECIST v1.1) for cohort1 and cohort2.
PFS2/PFS1(Progression Free Survival 2/Progression Free Survival 1) | Through study completion, an expected average of 1 year.
  For cohort3,the time to progression-free survival during the substudy (PFS2) exceeds the documented time to disease progression-free survival during the last treatment prior to substudy entry (PFS1) by at least 35% (ie, PFS2/PFS1≥1.3) or, if PFS1 is not evaluable, time to progressive disease exceeds 6 months.

SECONDARY OUTCOMES:
Progression Free Survival(PFS) | From treatment administration up to a maximum duration of 18 months
  The time from the beginning of the patient's treatment to the disease progression or death for any reason.Based on RECIST criteria v1.1
Overall Survival(OS) | From treatment administration up to a maximum duration of 18 months
  Time from start of treatment to death due to any cause.
Disease Control Rate (DCR) | From treatment administration up to a maximum duration of 18 months
  The proportion of subjects with complete response (CR) and partial response (PR) and stable disease (SD) in total subjects 12 months after the last subject participating in.
Time to response (TTR) | From treatment administration up to a maximum duration of 18 months.
  TTR (per RECIST 1.1) is defined as the time from the starting date of study drug to the first time complete response (CR) or partial response (PR) 12 months after the last subject participating in.
Percentage of Participants With Adverse Events (AEs) | From treatment administration up to a maximum duration of 18 months.
  Number of participants with adverse effects of treatment. Frequency and severity of adverse effects of treatment as assessed by NCI CTCAE v5.0.

CONTACTS AND LOCATIONS:
Locations (1):
- Tianjin Medical Unversity Second Hospital, Tianjin, Tianjin Municipality, China

IPD SHARING:
Plan to Share IPD: No